CLINICAL TRIAL: NCT06282328
Title: HIV HOspital TEsting: Bringing the Hidden to Light in the Hospital Setting: A Monocentric Observational Cross-Sectional Study
Brief Title: HIV HOspital TEsting: Bringing the Hidden to Light in the Hospital Setting
Acronym: HIV-HOTE
Status: Completed | Type: Observational
Sponsor: Castagna Antonella (Other)
Responsible Party: Sponsor-Investigator, Castagna Antonella, Prof, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: CET 26-2024
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hiv; HIV Infections; AIDS
Keywords: HIV; Screening; HIV Testing; HIV Screening; HIV Indicator Conditions; HIV IC
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — HIV Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HIV test — Bedside rapid capillary HIV test

SUMMARY:
This study aims to evaluate the prevalence of previously undiagnosed HIV infection in the hospital setting (across various medical or surgical departments) among individuals exhibiting at least one HIV indicator condition (HIV-IC) and/or engaging in risky behaviors.

This is a cross-sectional, single-center study with additional procedures. Data collection will involve clinical and laboratory data from individuals with at least one HIV-IC and/or behavioral risk factor for HIV infection admitted to the San Raffaele Hospital in Milan for any reason.

The overall study duration is 24 months, with recruitment lasting 20 months. Individuals will be actively recruited from various medical or surgical units of the hospital. After obtaining informed consent, clinical and laboratory information related to the study will be collected, along with specific blood samples. The presence of at least one HIV-IC will be determined using available clinical, radiological, and laboratory parameters during hospitalization.

Following informed consent, hospitalized individuals will complete a paper questionnaire, aimed at identifying behavioral risk factors for HIV infection. If at least one HIV-IC or behavioral risk factor is present, the person will be eligible for inclusion in the clinical study, and a rapid capillary HIV test will be conducted bedside.

In case of a positive rapid capillary HIV test result, antigen/antibody testing and Western Blot for HIV confirmation will be performed on venous blood samples on the same day.

DETAILED DESCRIPTION:
Study Objective:

This study aims to evaluate the prevalence of previously undiagnosed HIV infection in the hospital setting (across various medical or surgical departments) among individuals exhibiting at least one HIV indicator condition (HIV-IC) and/or engaging in risky behaviors.

Study Design:

This is a cross-sectional, single-center study with additional procedures. Data collection will involve clinical and laboratory data from individuals with at least one HIV-IC and/or behavioral risk factor for HIV infection admitted to the San Raffaele Hospital in Milan for any reason.

Study Duration:

The overall study duration is 24 months, with recruitment lasting 20 months, data extraction and review taking 2 months, statistical analysis requiring 1 month, and result writing taking 1 month.

Study Procedure:

Individuals will be actively recruited from various medical or surgical units of the hospital. After obtaining informed consent, clinical and laboratory information related to the study will be collected, along with specific blood samples. The presence of at least one HIV-IC will be determined using available clinical, radiological, and laboratory parameters during hospitalization.

Additional Procedures or Analyses:

* Following informed consent, hospitalized individuals will complete a paper questionnaire, aimed at identifying behavioral risk factors for HIV infection. If at least one HIV-IC or behavioral risk factor is present, the person will be eligible for inclusion in the clinical study, and a rapid capillary HIV test will be conducted bedside.
* In case of a positive rapid capillary HIV test result, antigen/antibody testing (using Cobas 6800®) and Western Blot for HIV confirmation will be performed on venous blood samples on the same day at the San Raffaele Hospital virology laboratory in Milan.
* If HIV infection is confirmed, an infectious disease specialist will assess the patient within 48 hours of diagnosis and request viral load determination (HIV-RNA), CD4+ lymphocyte count. The individual will also be directed to follow-up care at the Infectious Diseases Unit of San Raffaele Hospital, with subsequent linkage to care and start of antiretroviral therapy (ART), according to clinical practice.
* If the capillary HIV test result is negative, the patient will be informed of the negative result.

ELIGIBILITY:
Inclusion Criteria:

* Individuals admitted to various Units of IRCCS San Raffaele Hospital.
* Individuals aged 14 years or older.
* Individuals meeting at least one of the following criteria:

  * Presence of at least one HIV-IC.
  * Presence of at least one behavioral risk factors for HIV infection.
* Individuals providing specific written informed consent for the study, or minors whose parents or legal guardians provide specific written informed consent for the study.

Exclusion Criteria:

* Individuals not providing specific written informed consent for the study.
* Individuals with previously known HIV infection.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals admitted to various Units of San Raffaele Hospital (medical or surgical area).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of HIV infection | Month 20
  The primary objective of the study is to estimate the prevalence of previously unknown HIV infection (new HIV infection) in the hospital setting among individuals exhibiting at least one HIV indicator condition (HIV-IC) and/or with presence of behavioral risk factors

SECONDARY OUTCOMES:
Number of HIV-IC | Month 20
  The number/categories of HIV-IC will be assessed. HIV-IC will be defined according to ECDC HIV-IC guidelines
Number of Behavioral Risk Factors | Month 20
  The number/type of behavioral risk factors will be assessed. Presence of behavioral risk factors for HIV infection will be evaluated by means of a questionnaire designed for the trial
CD4+ lymphocytes | Month 20
  CD4+ lymphocytes (cells/microL) will be assessed among people with HIV infection at time of diagnosis
HIV-RNA | Month 20
  HIV-RNA levels (copies/mL) will be assessed among people with HIV infection at time of diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Nozza, MD, Principal Investigator — Vita-Salute San Raffaele University
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy